CLINICAL TRIAL: NCT04724538
Title: Inhalation Low Dose Radionuclide Therapy in Comprehensive Treatment of COVID-19 Viral Pneumonia
Brief Title: Inhalation Low Dose Radionuclide Therapy in Treatment COVID-19
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Medical Research Radiological Centre of the Ministry of Health of Russia (Other)
Responsible Party: Principal Investigator, Andrey Kaprin, general director of the National Medical Research Radiological Centre of the Ministry of Health of Russia, National Medical Research Radiological Centre of the Ministry of Health of Russia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RNT COVID-19
Record Dates: First submitted 2020-12-29; First posted 2021-01-26 (Actual); Results first posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Covid19; Pneumonia, Viral
Keywords: COVID-19; viral pneumonia; radionuclide therapy
MeSH Terms: conditions — COVID-19; Pneumonia, Viral

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy volunteers (Experimental): CT-scans for exclusion of pneumonia. Accumulated absorbed dose calculation of volunteers' lungs after inhalation of 99mTc-pertechnetate aerosol from commercial gas generator which was loaded by 833 MBq of 99mTc-pertechnetate.
  Interventions: Radiation: 99mTc-pertechnetate aerosol
- Patient with COVID-19 pneumonia (Experimental): Inhalation of 99mTc-pertechnetate aerosol from commercial gas generator which was loaded by 4165 MBq of 99mTc-pertechnetate. CT scans a day before, 7 and 14 days after inhalation procedure. Blood tests a day before, 1, 3 and 7 days after inhalation procedure.
  Interventions: Drug: 99mTc-pertechnetate aerosol
- Patient with COVID-19 pneumonia without intervention (No Intervention): Blood tests at 1, 3 and 7 days.

INTERVENTIONS:
Radiation: 99mTc-pertechnetate aerosol — 99mTc-pertechnetate is 99mTc-labeled carbon ultrafine aerosol
  Arms: Healthy volunteers
Drug: 99mTc-pertechnetate aerosol — 99mTc-pertechnetate is 99mTc-labeled carbon ultrafine aerosol
  Arms: Patient with COVID-19 pneumonia

SUMMARY:
Coronavirus disease (COVID-19) is a pandemic of unprecedented proportions with an exponential increase in incidence. Airway epithelium infection caused by coronavirus (SARS-CoV-2) triggers a cascade of difficult-to-control reactions, a so-called "cytokine storm". In contrast to the previously used method of external beam radiation therapy for patients at high risk of a cytokine storm, in present study a different dose delivery mechanism through inhalation of 99mTc-labeled carbon ultrafine aerosol obtained from a TechnegasPlus generator is used. By utilizing anthropometric phantoms the dosimetric characteristics of the applied technique and obtained the coefficients of the transition from the count rate over the area of interest to the activity contained in this area (in kBq) were studied. By observing a group of healthy volunteers after inhalation of 99mTc-labeled carbon ultrafine aerosol, the accumulated dose in the human lungs under internal irradiation of 99mTc was determined. A novel technique has been developed and the possibility of using inhaled low-dose radionuclide therapy in the complex treatment of patients with COVID-19 - associated pneumonia has been studied. As a result, a significant improvement of hematological parameters in the group of patients after inhalation of 99mTc-labeled carbon ultrafine aerosol as compared to the control group is expected.

ELIGIBILITY:
Inclusion Criteria:

1. Positive SARS-Cov-2 polymerase chain reaction (PCR)
2. CT confirmed pneumonia
3. Men and non-pregnant women ≥ 18 y/o with early laboratory signs of cytokine storm
4. Men and non-pregnant women <65 y/o and/or with early laboratory signs of cytokine storm
5. Informed consent obtained for participation

Exclusion Criteria:

1. Age ≤ 18
2. Severe course of COVID-19
3. Pregnant or breast-feeding females
4. Severe concomitant pathology
5. Previous and/or present treatment of oncology disease (e.g. immunotherapy)
6. Autoimmune diseases, severe cardiac disease, bone marrow and/or visceral transplantation
7. Surgical treatment and/or radiotherapy of chest pathology
8. Treatment with specific antiviral and anticytokine agents a day before inhalation procedure
9. Absence of informed consent obtained for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-03-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- P. Hertsen Moscow Oncology Research Institute, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patient With COVID-19 Pneumonia | Patient With COVID-19 Pneumonia Without Intervention
Started | 11 | 14
Completed | 11 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient With COVID-19 Pneumonia | Patient With COVID-19 Pneumonia Without Intervention | Total
Number analyzed (Participants) | 11 | 14 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 4 | 8 | 12
Age, Continuous [Mean (Full Range); unit: Years] | 54.3 [45 to 77] | 59.9 [53 to 67] | 57.5 [45 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 7 | 9 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 14 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Russia | 11 | 14 | 25

OUTCOME MEASURES:

1. Primary Outcome: Count of White Blood Cells (WBC) After 99mTc-pertechnetate Aerosol Inhalation for Adverse Events Monitoring as Evaluation Safety of This Procedure in Patients With COVID-19 Viral Pneumonia.
Description: Patients with COVID-19 viral pneumonia were observed for safety after administration of 99mTc-pertechnetate aerosol inhalation, and followed up at 1, 3, 7 days after inhalation. Patients did blood test to observe for abnormalities in clinical parameters and compare to baseline results as assessed by CTCAE v5.0. These tests were also performed in patients with COVID-19 viral pneumonia receiving standard treatment. The results were compared between the two groups.
Time Frame: Days 1, 3 and 7 after inhalation
Population: Count of white blood cells (WBC)
Measure: Mean (Standard Deviation); unit: x 1000 cells/microL
Arm/Group | Patient With COVID-19 Pneumonia | Patient With COVID-19 Pneumonia Without Intervention
Number analyzed (Participants) | 11 | 14
x 1000 cells/microL
  WBC - 1st day | 11.2 (4.5) | 9.8 (6.1)
  WBC - 3rd day | 9.7 (1.9) | 8.7 (6.3)
  WBC - 7th day | 8.8 (3.6) | 9.3 (2.1)

2. Primary Outcome: Count of Red Blood Cells (RBC) After 99mTc-pertechnetate Aerosol Inhalation for Adverse Events Monitoring as Evaluation Safety of This Procedure in Patients With COVID-19 Viral Pneumonia.
Description: as for outcome 1
Time Frame: Days 1, 3 and 7 after inhalation
Population: Count of red blood cells (RBC)
Measure: Mean (Standard Deviation); unit: x million cells/microL
Arm/Group | Patient With COVID-19 Pneumonia | Patient With COVID-19 Pneumonia Without Intervention
Number analyzed (Participants) | 11 | 14
x million cells/microL
  RBC - 1st day | 4.5 (0.6) | 4.5 (0.4)
  RBC - 3rd day | 4.3 (0.4) | 4.4 (0.5)
  RBC - 7th day | 4.2 (0.3) | 4.4 (0.2)

3. Primary Outcome: Hemoglobin Count (Hb) After 99mTc-pertechnetate Aerosol Inhalation for Adverse Events Monitoring as Evaluation Safety of This Procedure in Patients With COVID-19 Viral Pneumonia.
Description: as for outcome 1
Time Frame: Days 1, 3 and 7 after inhalation
Population: Hemoglobin count (Hb)
Measure: Mean (Standard Deviation); unit: gm/L
Arm/Group | Patient With COVID-19 Pneumonia | Patient With COVID-19 Pneumonia Without Intervention
Number analyzed (Participants) | 11 | 14
gm/L
  Hb - 1st day | 140.5 (20.7) | 132 (12.2)
  Hb - 3rd day | 137.5 (20.5) | 130.6 (13.2)
  Hb - 7th day | 135.3 (16.4) | 131 (14.4)

4. Primary Outcome: Percentage of Neutrophils (N) After 99mTc-pertechnetate Aerosol Inhalation for Adverse Events Monitoring as Evaluation Safety of This Procedure in Patients With COVID-19 Viral Pneumonia.
Description: as for outcome 1
Time Frame: Days 1, 3 and 7 after inhalation
Population: Percentage of neutrophils (N)
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Patient With COVID-19 Pneumonia | Patient With COVID-19 Pneumonia Without Intervention
Number analyzed (Participants) | 11 | 14
percentage
  Percentage of Neutrophils - 1st day | 76.3 (9.98) | 72.2 (10.4)
  Percentage of Neutrophils - 3rd day | 68.8 (10.7) | 72.2 (12.3)
  Percentage of Neutrophils - 7th day | 68.4 (9.3) | 71.5 (13.1)

5. Primary Outcome: Absolute Neutrophil Count (ANC) After 99mTc-pertechnetate Aerosol Inhalation for Adverse Events Monitoring as Evaluation Safety of This Procedure in Patients With COVID-19 Viral Pneumonia.
Description: as for outcome 1
Time Frame: Days 1, 3 and 7 after inhalation
Population: Absolute neutrophil count (ANC)
Measure: Mean (Standard Deviation); unit: x 1000 cells/microL
Arm/Group | Patient With COVID-19 Pneumonia | Patient With COVID-19 Pneumonia Without Intervention
Number analyzed (Participants) | 11 | 14
x 1000 cells/microL
  ANC - 1st day | 8.8 (4.5) | 7.4 (5.9)
  ANC - 3rd day | 6.8 (2.0) | 6.6 (6.1)
  ANC - 7th day | 6.2 (3.4) | 6.9 (2.9)

6. Primary Outcome: Absolute Lymphocyte Count (ALC) After 99mTc-pertechnetate Aerosol Inhalation for Adverse Events Monitoring as Evaluation Safety of This Procedure in Patients With COVID-19 Viral Pneumonia.
Description: as for outcome 1
Time Frame: Days 1, 3 and 7 after inhalation
Population: Absolute Lymphocyte Count (ALC)
Measure: Mean (Standard Deviation); unit: x 1000 cells/microL
Arm/Group | Patient With COVID-19 Pneumonia | Patient With COVID-19 Pneumonia Without Intervention
Number analyzed (Participants) | 11 | 14
x 1000 cells/microL
  ALC - 1st day | 1.6 (0.6) | 1.6 (0.7)
  ALC - 3rd day | 2.1 (0.9) | 1.4 (0.5)
  ALC - 7th day | 1.64 (0.5) | 1.73 (0.3)

7. Primary Outcome: Level of Lactate in the Blood After 99mTc-pertechnetate Aerosol Inhalation for Adverse Events Monitoring as Evaluation Safety of This Procedure in Patients With COVID-19 Viral Pneumonia.
Description: as for outcome 1
Time Frame: Days 1, 3 and 7 after inhalation
Population: Level of lactate in the blood
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Patient With COVID-19 Pneumonia | Patient With COVID-19 Pneumonia Without Intervention
Number analyzed (Participants) | 11 | 14
mmol/L
  Lactate - 1st day | 5 (1.9) | 4.11 (1.5)
  Lactate - 3rd day | 4.4 (1.4) | 4.6 (1.7)
  Lactate - 7th day | 4.28 (1.0) | 4.81 (1.9)

8. Primary Outcome: Level of D-dimer in Blood After 99mTc-pertechnetate Aerosol Inhalation for Adverse Events Monitoring as Evaluation Safety of This Procedure in Patients With COVID-19 Viral Pneumonia.
Description: as for outcome 1
Time Frame: Days 1, 3 and 7 after inhalation
Population: Level of D-dimer in blood
Measure: Mean (Standard Deviation); unit: ngm/mL
Arm/Group | Patient With COVID-19 Pneumonia | Patient With COVID-19 Pneumonia Without Intervention
Number analyzed (Participants) | 11 | 14
ngm/mL
  D-dimer - 1st day | 1737 (1172) | 1284 (1203)
  D-dimer - 3rd day | 843 (705) | 685 (579)
  D-dimer - 7th day | 383 (255) | 859 (693)

9. Secondary Outcome: Level of CD4+ T-cells in Blood After 99mTc-pertechnetate Aerosol Inhalation for Evaluation of Cellular Immune Response After This Procedure in Patients With COVID-19 Viral Pneumonia
Description: as for outcome 1
Time Frame: Days 1, 3 and 7 after inhalation
Population: Level of CD4+ T-cells in blood
Measure: Mean (Standard Deviation); unit: x 1000 cells/microL
Arm/Group | Patient With COVID-19 Pneumonia | Patient With COVID-19 Pneumonia Without Intervention
Number analyzed (Participants) | 11 | 14
x 1000 cells/microL
  CD4 - 1st day | 761 (365) | 614 (228)
  CD4 - 3rd day | 1100 (721) | 832 (546)
  CD4 - 7th day | 845 (447) | 718 (452)

10. Secondary Outcome: Level of NK-cells in Blood After 99mTc-pertechnetate Aerosol Inhalation for Evaluation of Cellular Immune Response After This Procedure in Patients With COVID-19 Viral Pneumonia
Description: as for outcome 1
Time Frame: Days 1, 3 and 7 after inhalation
Population: Level of NK-cells in blood
Measure: Mean (Standard Deviation); unit: x 1000 cells/microL
Arm/Group | Patient With COVID-19 Pneumonia | Patient With COVID-19 Pneumonia Without Intervention
Number analyzed (Participants) | 11 | 14
x 1000 cells/microL
  NK - 1st day | 153 (83) | 164 (72)
  NK - 3rd day | 188 (83) | 149 (77)
  NK - 7th day | 219 (92) | 181 (97)

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | Patient With COVID-19 Pneumonia | Patient With COVID-19 Pneumonia Without Intervention
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/14
Other Adverse Events (participants affected / at risk) | 0/11 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/38/NCT04724538/Prot_SAP_ICF_000.pdf